CLINICAL TRIAL: NCT05816538
Title: The Immune Response of Breast Cancer Patients Treated With Levobupivacaine Using Paravertebral or Superficial Chest Blocks
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rijeka (Other)
Responsible Party: Principal Investigator, Ivan Ivanovski, Principal investigator; Specialist in anesthesiology, reanimatology and intensive medicine, University of Rijeka
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2170-29-02/1-2
Record Dates: First submitted 2023-01-16; First posted 2023-04-18 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Paravertebral Block; Pectoralis and Serratus Plane Nerve Blocks; Breast Cancer; Immunologic Suppression; Levobupivacaine
Keywords: Breast Cancer; Levobupivacaine; Immunologic Suppression; Paravertebral block; Pectoralis and Serratus Plane Nerve Blocks
MeSH Terms: conditions — Breast Neoplasms | interventions — Anesthesia, General

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 PVB (Active Comparator): Group 1 will receive paravertebral block (PVB) as analgesia for breast surgery. PVB is a regional anesthetic technique applied at the thoracic (Th) level of Th2, Th3, and Th4 at a dose of 0.3ml/kg 0.5% levobupivacaine total, divided into levels. Block will be performed with ultrasound-guided in-plane technique and neurostimulation.
  Interventions: Procedure: Paravertebral nerve block (PVB); Device: Regional anesthetic technique with ultrasound guidance; Device: Regional anesthetic technique with peripheral nerve stimulation.; Drug: Levobupivacaine 0.5%; Procedure: General anesthesia
- Group 2 PECS (Experimental): Group 2 will receive Pectoralis and Serratus Plane Nerve blocks (PECS 2) as analgesia for breast surgery. PECS 2 block is a regional anesthetic technique applied in the space between the large and small pectoral muscles (10 ml of 0.5% levobupivacaine), and in the space between the small pectoralis muscle and the serratus anterior muscle (with 15 ml of 0.5% levobupivacaine). Block will be performed with ultrasound-guided in-plane technique and neurostimulation.
  Interventions: Procedure: Pectoralis and Serratus Plane Nerve Blocks (PECS 2); Device: Regional anesthetic technique with ultrasound guidance; Device: Regional anesthetic technique with peripheral nerve stimulation.; Drug: Levobupivacaine 0.5%; Procedure: General anesthesia

INTERVENTIONS:
Procedure: Paravertebral nerve block (PVB) — PVB is a regional anesthetic technique applied at the thoracic (Th) level of Th2, Th3, and Th4 at a dose of 0.3ml/kg 0.5% levobupivacaine total, divided into levels. Block will be performed with ultrasound-guided in-plane technique and neurostimulation.
  Arms: Group 1 PVB
Procedure: Pectoralis and Serratus Plane Nerve Blocks (PECS 2) — Pectoralis and Serratus Plane Nerve blocks (PECS 2) is a regional anesthetic technique applied in the space between the large and small pectoral muscles (10 ml of 0.5% levobupivacaine), and in the space between the small pectoralis muscle and the serratus anterior muscle (with 15 ml of 0.5% levobupivacaine). Block will be performed with ultrasound-guided in-plane technique and neurostimulation.
  Arms: Group 2 PECS
Device: Regional anesthetic technique with ultrasound guidance — The device that will be used is an ultrasound with an 8 Hz ultrasonic linear probe for both regional anesthetic techniques.
Device: Regional anesthetic technique with peripheral nerve stimulation. — The 22G neurostimulator needle (Stimuplex D®, B. Braun Melsungen AG)], and neurostimulator (Stimuplex HNS 12, B. Braun, Melsungen AG, Germany) will be used for both regional anesthesias.
Drug: Levobupivacaine 0.5% — Local anesthetic levobupivacaine 0.5% will be used for regional anesthetic technique with ultrasound guidance and peripheral nerve stimulation. For the paravertebral block at a dose of 0.3ml/kg total, applied at the thoracic (Th) level of Th2, Th3, and Th4 and divided into levels. For the PECS 2 block levobupivacaine 0.5% 10 ml will be applied in the space between the large and small pectoral muscles and 15 ml in the space between the small pectoralis muscle and the serratus anterior muscle.
Procedure: General anesthesia — In both groups for induction of general anesthesia we will use 1% propofol 2 - 2.5 mg/kg (10 mg/ml, Fresenius), sufentanil (Sufentanil® Altamedics) 0.2 μg / kg, rocuronium [Zemuron®, Schering - Plow] 0.8 mg/kg. We will use a laryngeal mask (I - gel supraglottic airway) of appropriate sizes for airway maintenance. All subjects will be ventilated by controlled mechanical ventilation with a volume of 8 ml/kg, a frequency of about 12 breaths per min with a mixture of oxygen and air in a 40: 60% ratio. Maintenance of anesthesia and sedation in group 1 will be performed with continuous infusion of 1% propofol (10 mg / ml, Fresenius) (25 - 150 mcg / kg / min.) and rocuronium [Zemuron®, Schering - Plow] 0.01 mg / kg / min per perfusor.

SUMMARY:
The use of regional anesthesia in breast surgery improves the postoperative outcome, reduces the development of infection, and weakens the perioperative immunosuppressive response associated with the response to surgical stress. The investigators hypothesize that the use of propofol / paravertebral anesthesia and analgesia will be accompanied by a decrease in serum proinflammatory cytokines and/or an increase in anti-inflammatory cytokines compared to propofol / PECS 2 anesthesia and analgesia. The research will be on 100 respondents divided into two groups. 0.5% levobupivacaine will be administered to both groups. Serum concentrations of pro- and anti-inflammatory cytokines, and lymphocyte subpopulations 1h before, 24h, and 48h after surgery will be measured. The investigators aim to compare the effect of propofol / paravertebral and propofol / PECS 2 anesthesia and analgesia on serum perioperative values of pro-inflammatory and anti-inflammatory cytokines to standardize protocols and apply the best method of perioperative analgesia in breast cancer surgery.

DETAILED DESCRIPTION:
Introduction

The human immune system is extremely adaptable and complex. The immune response in the body is often a defense against tumors or infection and maintenance of homeostasis. It includes specific (acquired) and nonspecific (innate) immunity. The immune system is known to be shaped by a complex network of cytokines; interleukins (IL), interferons (IFN), tumor necrosis factor [Eng. Tumor necrosis factor (TNF)] etc. Tumor cells respond differently to cytokines. Certain cytokines stimulate immune reactions and are called pro-inflammatory, while others inhibit the immune system response and are called anti-inflammatory. In previous studies, Il-1, Il-6, TNFα, and IL-10 are common indicators of inflammatory changes in cancer. IL-6 is a potent proinflammatory cytokine with multiple mechanisms of antitumor activity. TNFα stimulates the production of other proinflammatory factors and proteases. IL-10 inhibits the production of pro-inflammatory cytokines.

Surgery and anesthesia change the activity of the immune system quickly and through various processes. Pain, fear, medications, inhalation anesthetics, opioids, tissue injury, blood transfusions, increased stress, and infection activate the immune system during the perioperative period by suppressing the adaptive immune response or enhancing the immune response.

Breast cancer is the most common malignancy in women, second only to lung cancer in mortality. Breast cancer surgery is the primary and most effective treatment, with special emphasis on the minimal release of tumor cells into the vascular and lymphatic systems. Whether the release of tumor cells will result in clinical metastases depends primarily on the balance between antimetastatic immune activity and the ability of the tumor to metastasize to other tissues.

Regional anesthesia is a technique in which the application of a local anesthetic near a nerve or spinal cord inhibits the sensation, pain, and motor stimulation of one region of the body. Applied local anesthetics thus prevent the endocrine-metabolic response to stress. Many studies have shown that the use of neuraxial (spinal and epidural) and perineuroaxial paravertebral block (PVB) regional anesthesia in breast surgery [(propofol / paravertebral block anesthesia - analgesia)] improve postoperative outcome and reduce the development of perioperative immunosuppressive response associated with surgical stress.

A paravertebral block is applied to the wedge-shaped anatomical space located bilaterally paravertebral, between the parietal pleura anteriorly; vertebrae, and intervertebral discs medially; and the upper transverse rib ligament posteriorly. Pectoralis and serratus plane nerve blocks 1 and 2 (PECS 1 and 2) are newer regional anesthesia techniques in which a local anesthetic is administered between the pectoral muscle sheets. Recent research has shown that the use of PECS 2 in breast cancer surgery has the same perioperative analgesic effect as a paravertebral block, with fewer side effects. Although it has been proven that it is the blocks of these nerves that achieve satisfactory analgesia in breast surgery, their influence on the perioperative immune response has not yet been proven, nor has a comparison of the body's immune response to surgical stimulation with PECS 2 and PVB.

Participants

In the prospective, randomized, monocentric study, the investigators will perform a study on 100 participants, divided into two groups, or 50 participants per group. In Group 1 propofol / paravertebral anesthesia and analgesia will be used; in Group 2 the investigators will use propofol / PECS 2 anesthesia and analgesia. The investigators will include women scheduled for quadrantectomy with equilateral axillary lymphadenectomy, anesthesia preoperative status (American Society of Anesthesiologists (ASA)) 1 and 2, aged 18 to 65 years. Exclusive criteria are patient rejection, ASA> 3, contraindication for local anesthetic, contraindications for planned regional anesthesia and analgesia, immunosuppressive therapy including corticosteroids, acute infection, history of chronic opioid use, presence of autoimmune disease, obesity (defined as body mass index BMI greater than 29.9 kg/m2).

Research plan

The research will be conducted at the Clinical Hospital Center Rijeka, Department of Anesthesiology, Reanimation and Intensive Medicine, the Surgery Department, and the Department of Physiology, Immunology, and Pathophysiology at the Faculty of Medicine, University of Rijeka. The devices that will be used are ultrasound (8 Hz ultrasonic linear probe), neurostimulator needle [22G (Stimuplex D®, B. Braun Melsungen AG)], neurostimulator (Stimuplex HNS 12, B. Braun, Melsungen AG, Germany), a bispectral index monitoring device (BIS A-2000 BIS monitor, Aspect Medical Systems, Newton, MA, USA), perfusor (B. Braun's Perfusor®), enzyme-linked immunosorbent assay (ELISA), flow cytometry device (FACSCalibur, Becton Dickinson, San Jose, CA, USA).

The randomization schedule will be implemented by a computer-free randomization service (Urbaniak, GC, & Plous, S. (2013) Research Randomizer (Version 4.0)). Retrieved May 20, 2021, from http: // www. randomizer.org. Standard preoperative preparation and supervision will be performed in the ward and the pre-and post-anesthesia units. The first blood sample will be taken to all participants 1 hour before surgery on arrival at the above unit. In Group 1 the investigators will apply PVB at the thoracic (Th) level of Th2, Th3, and Th4 at a dose of 0.3ml/kg 0.5% levobupivacaine total, divided into levels. In Group 2 the investigators will apply PECS 2 block with 10 ml of 0.5% levobupivacaine in the space between the large and small pectoral muscles, and 15 ml in the space between the small pectoralis muscle and the serratus anterior muscle. Both blocks will be performed with ultrasound-guided in-plane technique and neurostimulation, as described in the literature. In both groups for induction of general anesthesia, the investigators will use 1% propofol 2 - 2.5 mg/kg (10 mg/ml, Fresenius), sufentanil (Sufentanil® Altamedics) 0.2 μg / kg, rocuronium [Zemuron®, Schering - Plow] 0.8 mg/kg. The investigators will use a laryngeal mask (I - gel supraglottic airway) of appropriate sizes for airway maintenance. All subjects will be ventilated by controlled mechanical ventilation with a volume of 8 ml/kg, a frequency of about 12 breaths per min with a mixture of oxygen and air in a 40: 60% ratio. Maintenance of anesthesia and sedation in group 1 will be performed with continuous infusion of 1% propofol (10 mg/ml, Fresenius) (25 - 150 mcg/kg/min) and rocuronium [Zemuron®, Schering - Plow] 0.01 mg/kg/min via perfusor. After induction, mean arterial pressure, heart rate, oxygen saturation, and BIS values will be recorded every five minutes for the duration of the operation. Continuous infusion of 1% propofol (10 mg/ml, Fresenius) will be adjusted according to the target values of BIS devices in the range of 45 to 55.

At the end of the operation, the investigators will wake up the participants from anesthesia. Postoperatively, participants will be monitored in a post-anesthesia care unit (PACU) room where vital parameters (ECG, non-invasive blood pressure measurement, and saturation) and visual analgesic scale (VAS) [from 0 (no pain) to 10 (worst imaginable pain) according to Rawal will be notified. If pain with VAS> 3 is present, participants will receive diclofenac sodium (Voltaren®, Pliva) 75 mg i.v. in 100 ml of saline for 15min. If pain with VAS ≥ 6 is present, a combination of diclofenac sodium (Voltaren®, Pliva) 75 mg i.v. and tramal (Tramal® Stada) 100 mg in 500 ml saline will be obtained. In case of nausea and vomiting as assessed on a three-point scale (0 = no nausea and vomiting; 1 = nausea, no vomiting; 2 = vomiting with or without nausea) thietylperazine (Torecan®, Krka) will be administered in a dose of 0.1 mg/kg on a scale ≥1. If all vital parameters are satisfactory and there are no complications, the participants will be referred to the department after two hours postoperatively. There, non-invasive hemodynamic monitoring (pressure, ECG, heart rate, saturation) will be performed until the block resolution. During the first 24 hours, the recovery of patients will be monitored and VAS will be assessed every 3 hours. Appropriate analgesic measures (non-steroidal anti-inflammatory drugs or opioid analgesics) will be performed based on VAS values.

Venous blood samples will be collected 24 and 48 hours after surgery. All samples will be delivered to the laboratory on the same day where they will be processed and stored at -20 Cs until analysis. According to the manufacturer's instructions, serum concentrations of pro-inflammatory cytokines Il-1, Il-6, TNFα, and anti-inflammatory cytokine IL-10 will be analyzed using an ELISA test. Subpopulations of T lymphocytes (helper and cytotoxic), B lymphocytes, NK, and NKT cells will be analyzed and determined from the samples by flow cytometry. Serum subpopulations of Treg (FITC-CD4, APC-CD25, and PE-Foxp3 positive) in serum will also be determined according to the manufacturer's instructions.

Statistics

The group size was obtained by power analysis. Using Fisher's exact test, according to the paper by Deegan CA, Murray D, Doran P, et al. Anesthetic technique and the cytokine and matrix metalloproteinase response to primary breast cancer surgery. Reg Anesth. Pain Med. 2010; 35: 490-5; the expected difference in the share of interleukin level increase of at least 25% (expected increase in group 1 of 30% and group 2 of 5%) is assumed. For a test power of 85%, a significance level of α = 0.05, and an equal number of subjects in groups, at least 45 subjects per group should be included in the study. Power analysis was performed using MedCalcStatistical Software version 19.0.3 (MedCalc Software, Ostend, Belgium; https://www.medcalc.org; 2019) and G * Power for Windows version 3.1.9.2.

IBM SPSS Statistics, version 21.0 (www.spss.com) will be used in the data analysis.

The data will be presented in tables and graphs. An analysis of the normality of data distribution (Kolmogorov-Smirnov test) will be made, and according to the obtained results, appropriate data display methods and parametric and/or non-parametric statistical methods will be applied. Quantitative data will be presented through ranges, arithmetic means, and standard deviations i.e., median and interquartile ranges in cases of nonparametric distribution. Category data will be presented through absolute frequencies and associated shares.

Differences between individual measurements will be analyzed by observing the variance for repeated measurements, i.e. the Friedman test. Differences in individual measurement times will be analyzed by the independent t-test or the Mann-Whitney U test. Differences in categorical values will be analyzed by Fisher's exact test. An appropriate regression model will assess the effect of selected clinical variables on differences between study groups. All P values less than 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* quadrantectomy with equilateral axillary lymphadenectomy
* anesthesia preoperative status (American Society of Anesthesiologists (ASA)) 1 and 2

Exclusion Criteria:

* patient rejection
* ASA> 3
* contraindication for local anesthetic
* contraindications for planned regional anesthesia and analgesia
* immunosuppressive therapy including corticosteroids
* acute infection
* history of chronic opioid use
* presence of autoimmune disease
* obese definite body mass index BMI) greater than 29.9 kg/m2

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-18 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in measured serum cytokines using an ELISA test after PVB. | 1 hour before intervention to 48 hours after surgery
  Venous blood samples will be collected 1 hour before and 24 and 48 hours after surgery. Serum concentrations in picogram per milliliter of pro-inflammatory cytokines Il-1, Il-6, TNFα, and anti-inflammatory cytokine IL-10 will be analyzed using an ELISA test according to the manufacturer's instructions.
Change in measured serum cytokines using an ELISA test after PECS 2 block. | 1 hour before intervention to 48 hours after surgery
  Venous blood samples will be collected 1 hour before and 24 and 48 hours after surgery. Serum concentrations picogram per milliliter of pro-inflammatory cytokines Il-1, Il-6, TNFα, and anti-inflammatory cytokine IL-10 will be analyzed using an ELISA test according to the manufacturer's instructions.
Change in cell number of individual lymphocyte subpopulations determined by flow cytometry technique (FACSCalibur) after PVB application. | 1 hour before intervention to 48 hours after surgery
  Venous blood samples will be collected 1 hour before and 24 and 48 hours after surgery. Peripheral blood leukocytes (PBL) will be isolated using a fluorescence-activated single-cell sorting flow cytometry technique on the FACSCalibur Flow Cytometer machine. Flow cytometry is a laser-based technique that detects and analyzes the chemical and physical characteristics of cells or particles. Individual lymphocyte subpopulations: T lymphocytes (helper and cytotoxic), B lymphocytes, NK, Treg (FITC-CD4, APC-CD25, and PE-Foxp3 positive), and NKT cells will be analyzed and determined according to the manufacturer's instructions using specific cell marker antibodies. After gating density plots the results will be presented in the number of cells in a cubic millimeter of blood and compared using scatter graphs.
Change in cell number of individual lymphocyte subpopulations determined by flow cytometry technique (FACSCalibur) after PECS 2 block application. | 1 hour before intervention to 48 hours after surgery
  Venous blood samples will be collected 1 hour before and 24 and 48 hours after surgery. Peripheral blood leukocytes (PBL) will be isolated using a fluorescence-activated single-cell sorting flow cytometry technique on the FACSCalibur Flow Cytometer machine. Flow cytometry is a laser-based technique that detects and analyzes the chemical and physical characteristics of cells or particles. Individual lymphocyte subpopulations: T lymphocytes (helper and cytotoxic), B lymphocytes, NK, Treg (FITC-CD4, APC-CD25, and PE-Foxp3 positive), and NKT cells will be analyzed and determined according to the manufacturer's instructions using specific cell marker antibodies. After gating density plots the results will be presented in the number of cells in a cubic millimeter of blood and compared using scatter graphs.

SECONDARY OUTCOMES:
Duration of postoperative analgesia after PVB application measured using visual analgesic scale (VAS). | 24 postoperative hours
  Postoperatively the subjects will be monitored in a post-anesthesia care unit (PACU) room where visual analgesic scale (VAS) [from 0 (no pain) to 10 (worst imaginable pain) according to Rawal will be notified at arrival to PACU, 1 hour and 2 hours postoperatively. Then the participants will be transferred to the department where, during the first 24 hours, the VAS will be assessed every 3 hours.
Duration of postoperative analgesia after PECS 2 block application measured using visual analgesic scale (VAS). | 24 postoperative hours
  Postoperatively the subjects will be monitored in a post-anesthesia care unit (PACU) room where visual analgesic scale (VAS) [from 0 (no pain) to 10 (worst imaginable pain) according to Rawal will be notified at arrival to PACU, 1 hour and 2 hours postoperatively. Then the participants will be transferred to the department where, during the first 24 hours, the VAS will be assessed every 3 hours.
The total dosage of analgesics in the postoperative period after the PVB application. | 48 postoperative hours
  The investigators will measure the total dosage of non-steroidal anti-inflammatory drugs (in mg) or opioid (in mg) analgesics in the first 48 hours after the PVB application.
The total dosage of analgesics in the postoperative period after the PECS 2 block application. | 48 postoperative hours
  The investigators will measure the total dosage of non-steroidal anti-inflammatory drugs (in mg) or opioid (in mg) analgesics in the first 48 hours after the PECS 2 application.
Mean atrial pressure change after the PVB. | From time of intervention to 2 hours postoperatively
  Before induction, mean arterial pressure (in mmHg) will be recorded using standard perioperative noninvasive blood pressure measurements at the time of block application, 60 min after, and at the time of transfer to the operating room. After induction, mean arterial pressure values will be recorded every five minutes for the duration of the operation. Postoperatively, subjects will be monitored in a post-anesthesia room where mean arterial pressure will be monitored at arrival, 1 hour and 2 hours postoperatively.
Mean atrial pressure change after the PECS 2 block. | From time of intervention to 2 hours postoperatively
  Before induction, mean arterial pressure (in mmHg) will be recorded using standard perioperative noninvasive blood pressure measurements at the time of block application, 60 min after, and at the time of transfer to the operating room. After induction, mean arterial pressure values will be recorded every five minutes for the duration of the operation. Postoperatively, subjects will be monitored in a post-anesthesia room where mean arterial pressure will be monitored at arrival, 1 hour and 2 hours postoperatively.
Change in the volume compensation of colloids after the PVB. | From the time of intervention to 24 hours postoperatively
  Total preoperative crystalloids infusions in milliliters will be recorded at the time of transfer to the operating room. Total intraoperative colloid infusions will be recorded at the end of the operation, before transfer to the PACU. Total postoperative crystalloids infusions will be recorded in PACU at the transfer to the department and after the first 24 hours at the department. The investigators will compare the difference between the two groups.
Change in the volume compensation of colloids after the PECS2 block. | From the time of intervention to 24 hours postoperatively
  Total preoperative colloid infusions in milliliters will be recorded at the time of transfer to the operating room. Total intraoperative colloid infusions will be recorded at the end of the operation, before transfer to the PACU. Total postoperative colloid infusions will be recorded in PACU at the transfer to the department and after the first 24h at the department. The investigators will compare the difference between the two groups.
Changes in heart rate values after the PVB. | From the time of intervention to 2 hours postoperatively
  Before induction heart rate (in beats per minute) will be recorded using standard perioperative ECG monitoring at the time of block application, 60 min after, and at the time of transfer to the operating room. After induction, heart rate values will be recorded every five minutes for the duration of the operation. Postoperatively, subjects will be monitored in a post-anesthesia room where heart rate will be monitored at arrival, 1 hour and 2 hours postoperatively.
Changes in heart rate values after the PECS 2 block. | From the time of intervention to 2 hours postoperatively
  Before induction heart rate (in beats per minute) will be recorded standard perioperative ECG monitoring at the time of block application, 60 min after, and at the time of transfer to the operating room. After induction, heart rate values will be recorded every five minutes for the duration of the operation. Postoperatively, subjects will be monitored in a post-anesthesia room where heart rate will be monitored at arrival, 1 hour and 2 hours postoperatively.
Change in the perioperative need for vasoactive drugs after PVB. | From the time of intervention to 2 hours postoperatively
  Total perioperative vasoactive drug applications in milligrams will be recorded at the end of the operation and before the transfer to the department. The investigators will compare the difference between the two groups in vasoactive drug application.
Change in the perioperative need for vasoactive drugs after PECS 2 block. | From the time of intervention to 2 hours postoperatively
  Total perioperative vasoactive drug applications in milligrams will be recorded at the end of the operation and before the transfer to the department. The investigators will compare the difference between the two groups in vasoactive drug application.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Ivanovski, M.D., Principal Investigator — Faculty of Medicine, University of Rijeka
Locations (1):
- University hospital centre Rijeka, Rijeka, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salo M. Effects of anaesthesia and surgery on the immune response. Acta Anaesthesiol Scand. 1992 Apr;36(3):201-20. doi: 10.1111/j.1399-6576.1992.tb03452.x. PMID 1574967
- [Background] Desborough JP. The stress response to trauma and surgery. Br J Anaesth. 2000 Jul;85(1):109-17. doi: 10.1093/bja/85.1.109. No abstract available. PMID 10927999
- [Background] Rao VS, Dyer CE, Jameel JK, Drew PJ, Greenman J. Potential prognostic and therapeutic roles for cytokines in breast cancer (Review). Oncol Rep. 2006 Jan;15(1):179-85. doi: 10.3892/or.15.1.179. PMID 16328053
- [Background] Nicolini A, Carpi A, Rossi G. Cytokines in breast cancer. Cytokine Growth Factor Rev. 2006 Oct;17(5):325-37. doi: 10.1016/j.cytogfr.2006.07.002. Epub 2006 Aug 22. PMID 16931107
- [Background] Deegan CA, Murray D, Doran P, Moriarty DC, Sessler DI, Mascha E, Kavanagh BP, Buggy DJ. Anesthetic technique and the cytokine and matrix metalloproteinase response to primary breast cancer surgery. Reg Anesth Pain Med. 2010 Nov-Dec;35(6):490-5. doi: 10.1097/AAP.0b013e3181ef4d05. PMID 20975461
- [Background] Kumari N, Dwarakanath BS, Das A, Bhatt AN. Role of interleukin-6 in cancer progression and therapeutic resistance. Tumour Biol. 2016 Sep;37(9):11553-11572. doi: 10.1007/s13277-016-5098-7. Epub 2016 Jun 3. PMID 27260630
- [Background] Sethi G, Sung B, Aggarwal BB. TNF: a master switch for inflammation to cancer. Front Biosci. 2008 May 1;13:5094-107. doi: 10.2741/3066. PMID 18508572
- [Background] Segerstrom SC, Miller GE. Psychological stress and the human immune system: a meta-analytic study of 30 years of inquiry. Psychol Bull. 2004 Jul;130(4):601-30. doi: 10.1037/0033-2909.130.4.601. PMID 15250815
- [Background] Antoni MH, Lutgendorf SK, Cole SW, Dhabhar FS, Sephton SE, McDonald PG, Stefanek M, Sood AK. The influence of bio-behavioural factors on tumour biology: pathways and mechanisms. Nat Rev Cancer. 2006 Mar;6(3):240-8. doi: 10.1038/nrc1820. PMID 16498446
- [Background] Sacerdote P, Bianchi M, Gaspani L, Manfredi B, Maucione A, Terno G, Ammatuna M, Panerai AE. The effects of tramadol and morphine on immune responses and pain after surgery in cancer patients. Anesth Analg. 2000 Jun;90(6):1411-4. doi: 10.1097/00000539-200006000-00028. PMID 10825330
- [Background] Bendre MS, Gaddy-Kurten D, Mon-Foote T, Akel NS, Skinner RA, Nicholas RW, Suva LJ. Expression of interleukin 8 and not parathyroid hormone-related protein by human breast cancer cells correlates with bone metastasis in vivo. Cancer Res. 2002 Oct 1;62(19):5571-9. PMID 12359770
- [Background] Holmgren L, O'Reilly MS, Folkman J. Dormancy of micrometastases: balanced proliferation and apoptosis in the presence of angiogenesis suppression. Nat Med. 1995 Feb;1(2):149-53. doi: 10.1038/nm0295-149. PMID 7585012
- [Background] Tsuchiya Y, Sawada S, Yoshioka I, Ohashi Y, Matsuo M, Harimaya Y, Tsukada K, Saiki I. Increased surgical stress promotes tumor metastasis. Surgery. 2003 May;133(5):547-55. doi: 10.1067/msy.2003.141. PMID 12773983
- [Background] Brown DL, Ransom DM, Hall JA, Leicht CH, Schroeder DR, Offord KP. Regional anesthesia and local anesthetic-induced systemic toxicity: seizure frequency and accompanying cardiovascular changes. Anesth Analg. 1995 Aug;81(2):321-8. doi: 10.1097/00000539-199508000-00020. PMID 7618723
- [Background] Homburger JA, Meiler SE. Anesthesia drugs, immunity, and long-term outcome. Curr Opin Anaesthesiol. 2006 Aug;19(4):423-8. doi: 10.1097/01.aco.0000236143.61593.14. PMID 16829725
- [Background] Mrakovcic-Sutic I, Bacic D, Golubovic S, Bacic R, Marinovic M. Cross-talk between NKT and regulatory T cells (Tregs) in modulation of immune response in patients with colorectal cancer following different pain management techniques. Coll Antropol. 2011 Sep;35 Suppl 2:57-60. PMID 22220404
- [Background] Zura M, Kozmar A, Sakic K, Malenica B, Hrgovic Z. Effect of spinal and general anesthesia on serum concentration of pro-inflammatory and anti-inflammatory cytokines. Immunobiology. 2012 Jun;217(6):622-7. doi: 10.1016/j.imbio.2011.10.018. Epub 2011 Nov 3. PMID 22217966
- [Background] Karmakar MK. Thoracic paravertebral block. Anesthesiology. 2001 Sep;95(3):771-80. doi: 10.1097/00000542-200109000-00033. No abstract available. PMID 11575553
- [Background] Kulhari S, Bharti N, Bala I, Arora S, Singh G. Efficacy of pectoral nerve block versus thoracic paravertebral block for postoperative analgesia after radical mastectomy: a randomized controlled trial. Br J Anaesth. 2016 Sep;117(3):382-6. doi: 10.1093/bja/aew223. PMID 27543533
- [Background] Schnabel A, Reichl SU, Kranke P, Pogatzki-Zahn EM, Zahn PK. Efficacy and safety of paravertebral blocks in breast surgery: a meta-analysis of randomized controlled trials. Br J Anaesth. 2010 Dec;105(6):842-52. doi: 10.1093/bja/aeq265. Epub 2010 Oct 14. PMID 20947592
- [Background] Blanco R, Fajardo M, Parras Maldonado T. Ultrasound description of Pecs II (modified Pecs I): a novel approach to breast surgery. Rev Esp Anestesiol Reanim. 2012 Nov;59(9):470-5. doi: 10.1016/j.redar.2012.07.003. Epub 2012 Aug 29. PMID 22939099